CLINICAL TRIAL: NCT04736745
Title: A Phase Ib/II, Multicentre, Double-blind, Randomised, Placebo-controlled Dose Escalation and Dose Finding Study to Evaluate the Safety and Efficacy of IPN59011 in Improving the Appearance of Moderate to Severe Upper Facial Lines
Brief Title: Study to Evaluate the Safety and Efficacy of IPN59011 in Improving the Appearance of Moderate to Severe Upper Facial Lines.
Acronym: LONG-SET
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor terminated the study due to strategic considerations
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-FR-59011-001; 2019-003268-33 (EudraCT Number)
Record Dates: First submitted 2021-01-12; First posted 2021-02-03 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Moderate Upper Facial Lines; Severe Upper Facial Lines
MeSH Terms: interventions — abobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: For dose escalation part Sequential study model will be used. For the rest of the study parallel assignment will be used.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose escalation (Experimental): One single injection of study medication (IPN59011 or Placebo) will be injected locally. IPN59011 is injected in a dose-escalation manner.
  In total for this stage at least 40 subjects.
  Interventions: Biological: IPN59011; Drug: Placebo
- Dose ranging (Experimental): Up to two IPN59011dose(s) groups will be included in parallel groups versus Azzalure group and placebo group. One single injection of study medication will be injected locally into several sites.
  In total for this stage at least 70 subjects.
  Interventions: Biological: IPN59011; Biological: Azzalure; Drug: Placebo
- Additional dose ranging (Experimental): Dose-ranging for three additional placebo-controlled parallel groups. One single injection of study medication will be injected locally into several sites, concomitantly and non-concomitantly.
  In total for this stage at least 110 subjects.
  Interventions: Biological: IPN59011; Drug: Placebo
- Total dose for Upper Facial Lines (Experimental): One single injection of study medication will be injected locally into Upper Facial Lines.
  In total for this stage approximately 48 subjects.
  Interventions: Biological: IPN59011; Drug: Placebo

INTERVENTIONS:
Biological: IPN59011 — Powder and solvent for solution for injection
Biological: Azzalure — Powder for solution for injection
  Arms: Dose ranging
Drug: Placebo — Powder for solution for injection

SUMMARY:
The purpose of the protocol, is to assess the safety and efficacy profile of IPN59011 compared to a placebo. IPN59011 is expected to work longer than product already marketed in the treatment of subjects with moderate to severe facial wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study related procedures.
* Female and male subjects between 18 and 65 years of age, inclusive (for dose escalation females only)
* Moderate or severe (Grade 2 or 3) GL at maximum contraction at Baseline, as assessed by the ILA using a validated 4-point photographic scale.
* Moderate or severe (Grade 2 or 3) GL at maximum contraction at Baseline, as assessed by the SSA using a validated 4-point categorical scale.
* Moderate or severe (Grade 2 or 3) Forehead Lines (FHL) at maximum contraction and moderate to severe GL at maximum contraction at Baseline or moderate to severe (Grade 2 or 3) Lateral Canthal Lines (LCL) at maximum contraction (Stage as assessed by the ILA using a validated 4-point photographic scale).
* Moderate or severe (Grade 2 or 3) FHL at maximum contraction and moderate to severe GL at maximum contraction at Baseline and moderate to severe (Grade 2 or 3) LCL at maximum contraction (Stage as assessed by the ILA using a validated 4-point photographic scale).
* Moderate or severe (Grade 2 or 3) FHL at maximum contraction and moderate to severe GL maximum contraction at Baseline or moderate to severe (Grade 2 or 3) LCL at maximum contraction, as assessed by the by the SSA using a validated 4-point categorical scale.
* Moderate or severe (Grade 2 or 3) FHL at maximum contraction and moderate to severe GL maximum contraction at Baseline and moderate to severe (Grade 2 or 3) LCL at maximum contraction, as assessed by the by the SSA using a validated 4-point categorical scale.
* Dissatisfied or very dissatisfied (Grade 2 or 3) with their lines at Baseline, as assessed by the subject's level of satisfaction.
* A negative pregnancy test (for females of childbearing potential only). Non-childbearing potential is defined as postmenopausal for at least 1 year; surgical sterilisation at least 3 months before entering the study; or hysterectomy.
* Subject has both the time and the ability to complete the study and comply with study instructions.

Exclusion Criteria:

* Previous treatment with any Botox (BTX) serotype (for dose escalation at least) or any recent treatment (within the past 6 months prior to Baseline for the rest of the study) with any BTX serotype.
* Any prior treatment with permanent fillers in the upper face including the GL, FHL and LCL area.
* Any prior treatment with long lasting dermal fillers in the upper face including the GL area within the past 3 years and/or skin abrasions/resurfacing (whatever the interventional technic used) within the past 5 years, or photo rejuvenation or skin/vascular laser intervention within the 12 months prior to Baseline.
* Any planned facial cosmetic surgery during the study.
* A history of eyelid blepharoplasty or brow lift within the past 5 years.
* An inability to substantially reduce GL by physically spreading them apart or lack of capacity to frown.
* An active infection or other skin problems in the upper face including the GL, FHL and LCL area (e.g. acute acne lesions or ulcers).
* Use of concomitant therapy which, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study treatment, including medications affecting bleeding disorders (e.g. antiplatelet agents and/or anticoagulants given for treatment or prevention of cardiovascular/cerebrovascular diseases).
* Pregnant women, nursing women, premenopausal women or women of childbearing potential (i.e. not surgically sterile or 1 year postmenopausal) not willing to practice a highly effective form of contraception method at the beginning of the study, for the duration of the study and for a minimum of 12 weeks following last administration of study treatment. Highly effective methods of contraception are defined as methods of birth control which result in a low failure rate (less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, intrauterine devices, or vasectomised partner.
* Male subjects who are not vasectomised and who have female partners of childbearing potential and are not willing to use condoms with spermicide throughout study participation for a minimum of 12 weeks following initial double-blind administration of the treatment.
* Positive for hepatitis B antigen, or hepatitis C virus antibody, or for human immunodeficiency virus (HIV) or a diagnosis of acquired immunodeficiency syndrome.
* A history of drug or alcohol abuse.
* Use of any experimental device within 30 days or use of any treatment with an experimental drug within five times the documented terminal half-life of the respective drug or its metabolites or if the half life is unknown within 30 days prior to the start of the study (prior to Baseline) and during the conduct of the study.
* Clinically diagnosed significant anxiety disorder, or any other significant psychiatric disorder (e.g. depression) that might interfere with the subject's participation in the study.
* Use of medications that affect neuromuscular transmission, such as curare-like nondepolarising agents, lincosamides, polymyxins, anticholinesterases and aminoglycoside antibiotics, within the past 30 days prior to Baseline.
* A history of facial nerve palsy.
* Marked facial asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin.
* Known allergy or hypersensitivity to BTX, or any excipients of IPN59011 or Azzalure, or allergy to cow's milk protein.
* Any known medical condition that may put the subject at increased risk in regard to exposure to BoNT of any serotype (i.e. myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, etc.)
* The presence of any other condition (e.g. neuromuscular disorder or other disorder that could interfere with neuromuscular function), laboratory finding or circumstance that, in the judgment of the investigator, might increase the risk to the subject or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
* Any uncontrolled systemic disease or other significant medical condition considered as an exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Incidence of the Treatment-Emergent Adverse Events (TEAEs) at each dose for dose escalation | from baseline until the end of study (9 months)
Incidence of Serious Adverse Events (SAEs) at each dose for dose escalation | from baseline until the end of study (9 months)
Incidence of clinically significant Adverse Events (AEs) at each dose for dose escalation | from baseline until the end of study (9 months)
Incidence of AEs (or SAEs) leading to withdrawals and Adverse Events of Special Interest (AESIs) for dose escalation | from baseline until the end of study (9 months)
Presence of botulinum neurotoxin serotype A (BoNT-A) antibodies and IPN59011 antibodies and titres (binding and neutralizing) | from baseline until the end of study (9 months)
Response to treatment measured by the composite response of 2-grade improvement on investigator's live assessment (ILA) at maximum contraction. | Day 29
  ILA: a validated 4-point photographic scale to assess the severity and appearance of the GLs at maximum frown and at rest where 0 is "no lines are noticeable" and 3 is "lines are extremely pronounced".
Response to treatment measured by the composite response of 2-grade improvement on subject's self-assessment (SSA) at maximum contraction. | Day 29
  SSA: a validated 4-point categorical scale to assess the appearance of their Glabellar Lines (GLs) at maximum frown where 0 is "no wrinkles" and 3 is "severe wrinkles".

SECONDARY OUTCOMES:
Response to treatment as measured by the reduction of ≥2 grades on the ILA at maximum contraction | From the baseline to the end of the study (9 months)
Response to treatment as achieved by a score of "none" or "mild" as measured by the ILA at maximum contraction | From the baseline to the end of the study (9 months)
Response to treatment as achieved by a score of "none" or "mild" as measured by the ILA at rest | From the baseline to the end of the study (9 months)
Response to treatment as measured by the reduction of ≥2 grades on the SSA at maximum contraction | From the baseline to the end of the study (9 months)
Response to treatment as achieved by a score of "none" or "mild" as measured by the SSA at maximum contraction | From the baseline to the end of the study (9 months)
Response to treatment as achieved by a score of "very satisfied" or "satisfied" on the Subject Level of Satisfaction (SLS) | From the baseline to the end of the study (9 months)
Duration of treatment response based on ILA and SSA at maximum contraction | From the baseline to the end of the study (9 months)
Face-Q (overall satisfaction with facial appearance) for Upper Facial Lines (UFL) | Visits screening, Day 1, Day 15, Day 29, 3 months, 6 months, 9 months
Time to onset of treatment response based on subject diary cards to evaluate the appearance of their lines. | From Day 1 through Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Clinical Research Centre (CRS), Berlin, Germany

IPD SHARING:
Plan to Share IPD: No